CLINICAL TRIAL: NCT05454618
Title: U-DECIDE: The Decision To Enroll In Therapeutic Clinical Trials In A Pediatric Cancer Clinical Network
Brief Title: The Decision To Enroll In Therapeutic Clinical Trials In A Pediatric Cancer Clinical Network
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: U-DECIDE; NCI-2022-05119 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2022-06-15; First posted 2022-07-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: Parent; Pediatric Oncology Patients; Caregivers; Barriers to Enrollment on a Therapeutic Trial; Parent Navigator Program; Affiliate Network; Decision Making; Healthcare; Parent Engagement
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The focus of this study is to learn about the factors that parents consider when making a decision for their child to participate or not in a clinical treatment research study.

DETAILED DESCRIPTION:
Aim 1:

* To describe the sociodemographic characteristics of patients treated through the Affiliate network, including those that are eligible for a therapeutic treatment study as well as those that are not. This aim will be accomplished using a survey based on previously validated tools measuring demographics, social determinants of health, and material hardship.

Following consent, the study team research assistant will verbally administer survey #1 to each participant or email the unique electronic link for each participant to complete. If necessary, survey #1 may be administered at a later date mutually agreed upon by the interviewer and the participant. Survey #1 contains questions on race, ethnicity, family structure, marital status, household income, and education level of parents, as well as previously validated instruments assessing cumulative hardship through assessments of housing, food accessibility, and utilities. Address information on both participants and non-participants will also be collected.

Aim 2:

* To examine the associations between social determinants, decision-making factors, trial-related attitudes, and additional individual preferences among parents/LARs of newly diagnosed pediatric oncology patients in the Affiliate network and the decision to enroll or not enroll on a therapeutic clinical trial. This aim will be accomplished through a convergent mixed-method design and include an additional exploratory qualitative sub-aim assessing potential differences in interviews conducted by parent versus non-parent interviewers.

Aim 2a:

* Quantitatively explore the relationship between social determinants and individual preferences among parents/LARs and the decision to enroll on a therapeutic clinical trial.

Parents/LARs who meet inclusion criteria for Aim 1, and are eligible for a clinical trial, will be included for potential participation. Data collected will include a subset of data collected for Aim 1, as well as data from a second survey (survey #2) focused on decision making and clinical trial attitudes. Additional items assessed with survey #2 relate to clinical trial attitudes and pediatric research participation including measures assessing access, risks of enrollment, attitudinal barriers, financial and social concerns, as well as trust/mistrust. Following consent, the study team research assistant will verbally or electronically administer survey #2 to each participant. If eligibility for clinical trial enrollment is known at the time of administration of survey #1, survey #2 may be administered at the same time to eligible parents/LARs. Otherwise, parents/LARs of children who are eligible for a clinical trial will be asked to complete survey #2 once this eligibility is confirmed and at a time mutually agreed upon by the participant and the research assistant.

In addition to the data collected from participants as described above, data from the affiliate log, including provider described reasons for non-enrollment on a clinical trial as applicable, will be collected.

Aim 2b:

* Qualitatively determine the relationship between social determinants, decision- making factors, trial related attitudes among parents/LARs and the decision to enroll or not enroll on a therapeutic clinical trial.

A subset of parents/LARs of children eligible for clinical trial enrollment will be approached to participate in a semi-structured interview. Participants for this qualitative sample will include a group of parents/LARs who decided to enroll, as well as a group of parents/LARs who chose not to enroll their child on a clinical trial.

Interviews will be conducted in either English or Spanish by bilingual interviewers using a semi-structured interview guide. These interviews will explore parents/LARS' general feelings about medical research including reasons they would or would not want their child to be enrolled in a research study, as well as more in-depth questions regarding their own experience talking to their child's oncologist about the clinical trial and their decision-making process around enrollment. Interviews will be conducted over the phone or a video-conferencing program platform by a trained qualitative interviewer and audio-recorded

Sub-aim 2b:

* Qualitatively explore differences between parent/LAR individual preferences as expressed to parent interviewers compared to non-parent interviewers.

Participants for this qualitative sample will be purposefully selected to mirror the qualitative sample included in aim 2b. Semi-structured interviews will be conducted in English or Spanish by bilingual parent interviewers. These interviews will be conducted over the phone or a video-conferencing program platform and audio-recorded. Parent interviewers will receive the same qualitative interview training as non-parent interviewers. The first portion of the interview guide will match the one used in investigator-led interviews. Additional questions will be added to the parent-interviewer guide including questions that address the participants comfort discussing clinical trial enrollment with parent interviewers.

Aim 3:

* To assess acceptability and feasibility of a parent navigator program within the Affiliate network.

All parents who choose to enroll their child in a clinical trial will be eligible for enrollment in the parent navigator program. The aim is to recruit and train 1-2 parent navigators at each affiliate site. Parent navigators will be recruited and trained based on the established process for the parent mentor program at St. Jude. Recruitment and training will begin in year 1 and continue through year 4 of the study.

Newly diagnosed parents/LARs whose children are eligible for enrollment on a therapeutic clinical trial will be offered enrollment in the pilot intervention. Once enrolled, parent navigators will initiate contact with parents of newly diagnosed patients first through a phone call or text message. Newly diagnosed parents/LARs will be paired with navigators for 6 weeks. Two interactions are proposed: one within weeks 1-3 of diagnosis/enrollment and the second during weeks 4-6, however, the navigator will be available for additional interactions as necessary and will contact the newly diagnosed parent/LAR approximately every 10 days. During this period, interactions between parents and navigators will be focused on initial decision-making around clinical trial enrollment, concerns regarding the clinical trial, confusion around elements of the clinical trial, and referrals to aid in information exchange.

After initiating contact with a newly diagnosed parent/LAR, parent navigators will complete an encounter form including a baseline questionnaire of parent and patient data as well as potential barriers to clinical trial enrollment. Following completion of the six weeks of engagement, both the parent- navigator and the parent/LAR will be asked to complete a final questionnaire. The parent questionnaire will include items related to satisfaction with the program and adapted to focus on clinical trial enrollment, as well as a brief instrument previously validated to assess acceptability and navigators will complete a questionnaire assessing acceptability and feasibility of the program.

ELIGIBILITY:
Inclusion Criteria:

* All English or Spanish speaking parents/LARs of patients 0-18 years of age with newly diagnosed cancer in the Affiliate network.

Exclusion Criteria:

* Parents of children with relapsed or recurrent disease, or those with benign neoplasms.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All English or Spanish speaking parents/LARs of patients 0-18 years of age with newly diagnosed cancer in the Affiliate network.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic characteristics of patients treated through the Affiliate network | Day 1, or during a future contact (approximately 1 month)
  Sociodemographic information will be analyzed descriptively. Full home address data will be geocoded to generate area deprivation information for each participant. Cumulative hardship will be calculated using previously established measures and scoring.These scores will be analyzed descriptively. Exploratory comparative analysis will be done to determine if there are differences between the sub-group of patients eligible for clinical trial enrollment versus those who are not eligible.
The correlation between social determinants and individual preferences among parents/LARs and the decision to enroll on a therapeutic clinical trial. | Day 1, or during a future contact (approximately 2 months)
  Data collected from survey #1 for this subgroup of patients will be used to statistically describe the sociodemographic information for patients who are eligible to enroll on a clinical trial and comparative analysis will be conducted to examine differences and potential associations between the group of parents/LARs who do enroll their child on a clinical trial, and those who do not. Responses from survey #2 will be analyzed descriptively to provide an overall understanding of decision-making preferences and roles, as well as clinical trial attitudes amongst parents/LARs whose children are eligible for a clinical trial. Comparative analysis will be used to determine if there are differences in these individual preference items between the group of parents/LARs whose children do enroll on a clinical trial, and those who do not.
The correlation between social determinants, decision-making factors, trial related attitudes among parents/LARs and the decision to enroll or not enroll on a therapeutic clinical trial. | Approximately 3 months after enrollment
  Qualitative data from semi-structured interviews will be transcribed and formally analyzed using thematic content analysis.
Differences between parent/LAR individual preferences as expressed to parent interviewers compared to non-parent interviewers | Approximately 3 months after enrollment
  Qualitative data will be formally analyzed using thematic content analysis comparing data collected by parent interviewers to data collected by non-parent interviewers.
Acceptability of a parent navigator program in the Affiliate network | After initiation of the Parent Navigator Program approximately 4 years after start of study
  Acceptability: we will determine that the navigator program is acceptable if the median score on the acceptability scale is > 3.
  Likert scale 1-5 will be used (1=Completely disagree, 2=Disagree, 3=Neither, 4=Agree, 5=Completely agree)
Feasibility of a parent navigator program in the Affiliate network | After initiation of the Parent Navigator Program approximately 4 years after start of study
  Feasibility: we will determine that the navigator program is feasible if the median score on the feasibility scale is > 3.
  Likert scale 1-5 will be used (1=Completely disagree, 2=Disagree, 3=Neither, 4=Agree, 5=Completely agree)

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Graetz, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols